CLINICAL TRIAL: NCT01790893
Title: Intravitreal Aflibercept Injection for the Treatment of cHoroidAl Neovascularization seconDary to Presumed ocuLar Histoplasmosis syndromE.(the HANDLE Study)
Brief Title: Treatment for Presumed Ocular Histoplasmosis
Acronym: HANDLE
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: John Kitchens, MD (Other)
Responsible Party: Sponsor-Investigator, John Kitchens, MD, Sponsor-Investigator, Retina Associates of Kentucky
Organization: Retina Associates of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IND 117497
Record Dates: First submitted 2013-02-11; First posted 2013-02-13 (Estimated); Last update posted 2014-06-16 (Estimated); Status verified 2014-06

CONDITIONS: Ocular Histoplasmosis
Keywords: Histoplasmosis
MeSH Terms: conditions — Histoplasmosis | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- intravitreal aflibercept injection (Experimental): Group A -Monthly intravitreal aflibercept injection for 3 months (Baseline, Months 1 and 2), then mandatory every 2 months intravitreal aflibercept injection (Months 4,6, 8 and 10)for 12 months. Monthly visits with evaluations for as needed intravitreal aflibercept injection.
  .
  Interventions: Drug: aflibercept
- intravitreal aflibercept (Experimental): Group B- One intravitreal aflibercept injection at Baseline, then monthly visits with evaluations for as needed dosing of intravitreal aflibercept injection for 12 months.
  Interventions: Drug: aflibercept

INTERVENTIONS:
Drug: aflibercept

SUMMARY:
The purpose of this study is to monitor safety outcomes for patients being treated with intravitreal aflibercept injections for choroidal neovascularization secondary to Presumed Ocular Histoplasmosis Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Active choroidal neovascularization (CNV) secondary to presumed ocular histoplasmosis demonstrated by active leakage on fluorescein angiography with spectal domain OCT evidence of subretinal or intraretinal fluid or PED.
* Active CNV may also be defined as demonstrating active subretinal hemorrhage.
* ETDRS Best corrected visual acuity 20/20-20/320.
* willing and able to comply with all study clinic visits and study related procedures.
* Willing to use and practice more than one form of contraceptives during the 13 month study for male and female.
* Provide signed informed consent
* Able to understand and complete study related questionnaires

Exclusion Criteria:

* Under 18 years of age
* CNV due to other causes than Presumed Ocular Histoplasmosis
* Previous treatment in the study eye within 6 months prior to Day 1
* More than 5 Intravitreal injections of anti-VEGF therapy within previous 12 months
* Any clinical evidence of any other ocular condition other than Ocular histoplasmosis
* History of allergy to fluorescein
* Pregnant( or planning on becoming pregnant within the next 13 months) or breast feeding women
* Sexually Active Men or Women who are NOT willing to practice more than one form of contraceptives during the next 13 months.
* Anticipated or previous (within previous 3 months) systemic anti-VEGF therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-03; Primary Completion 2014-08 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
ocular and systemic adverse events | through Month 12
  The primary objective of the study is the incidence and severity of ocular and systemic adverse events through Month 12

SECONDARY OUTCOMES:
Visual acuity | Months 3, 6, 9 and 12
  * Mean change in BCVA from Baseline
  * Proportion of subjects gaining >5,10 and 15 letters
  * Proportion of subjects losing >5, 10 and 15 letters

OTHER OUTCOMES:
OCT changes | baseline to 12 months
  Mean change from baseline in central subfield thickness over time up to 12 months assessed on OCT

CONTACTS AND LOCATIONS:
Overall Officials: John W Kitchens, MD, Principal Investigator — Retina Associates of Kentucky
Locations (3):
- United States (3):
  - Southeast Retina, Augusta, Georgia
  - Retina Associates of Kentucky, Lexington, Kentucky
  - Cincinnati Eye Institute, Cincinnati, Ohio

REFERENCES:
- See also: Related Info — http://www.retinaky.com